CLINICAL TRIAL: NCT06489275
Title: Testing an Intervention to Promote Financial Wellness Among Adults With Psychiatric Disabilities
Brief Title: Building Financial Wellness Randomized Controlled Trial
Acronym: BFW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Collaborative Support Programs of New Jersey (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY2020-1566
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Mental Disorder
Keywords: Financial Wellness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: The intervention improves financial literacy by imparting knowledge, increasing self-awareness of spending habits, building on existing money management skills, and setting personally-meaningful financial goals. During the course of the 6-session intervention, participants learn to set and begin working toward attainable financial goals. Learning occurs in a context of acceptance and encouragement aimed at increasing participants' sense of control over their personal finances. For 3 months after class ends, monthly booster sessions are held.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subjects receive a brief intervention consisting of 6 financial literacy classes designed to improve their financial literacy and financial wellness, followed by 3 one-on-one booster sessions to reinforce learning and provide support.
  Interventions: Behavioral: Building Financial Wellness
- Services as Usual (Active Comparator): Subjects receive routine mental health care.
  Interventions: Other: Services as Usual

INTERVENTIONS:
Behavioral: Building Financial Wellness — In addition to receiving services as usual, subjects attend financial literacy classes and booster sessions.
  Arms: Intervention
Other: Services as Usual — Subjects continue to receive services as usual.
  Arms: Services as Usual

SUMMARY:
This study tests a psychosocial intervention to improve financial literacy and behaviors among adults with mental illnesses.

DETAILED DESCRIPTION:
This study is designed to test the effectiveness of a financial education curriculum, called Building Financial Wellness (BFW), in promoting financial literacy and reducing economic strain among adults with a mental health condition. The design involves random assignment of adults who are receiving mental health services to the intervention plus services as usual, versus services as usual alone. Assessments at baseline, two months post-baseline, and three months later collect data to test the null hypotheses of no difference between intervention and control conditions on outcome measures in the following domains using longitudinal mixed-effects random regression analyses: 1) financial well-being; 2) financial strain; 3) financial capability; 4) financial self-sufficiency; and 5) financial literacy.

ELIGIBILITY:
Inclusion Criteria:

* age 18+
* access to computer, tablet or smart phone and an internet connection suitable for using Zoom
* receiving services and/or supports for a diagnosed mental health disorder
* ability to understand spoken English
* interest in learning money management skills.

Exclusion Criteria:

* Cognitive impairment preventing informed consent
* Unable to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Financial Wellness | study entry (pre-intervention), immediate post-intervention, 3 months post-intervention]
  The Consumer Financial Protection Bureau's Financial Well-Being Scale consists of 10-items and assesses the extent to which a person's financial status and capability provide them with security and freedom of choice. Respondents rate each item using a 5-point Likert scale ranging from "not at all" to "completely." Responses are coded 0-4 and summed for a total score potentially ranging from 0 to 40 with higher scores indicating greater financial well-being.

SECONDARY OUTCOMES:
Change in Financial Strain | study entry (pre-intervention), immediate post-intervention, 3 months post-intervention]
  The Financial Strain Questionnaire measures the level of distress associated with one's finances. This scale consists of 9-items and uses a 3-point Likert scale ranging from "no difficulty" to "great difficulty". Responses are coded 1-3 and summed for a total score potentially ranging from 9-27, with higher scores indicating greater financial strain.
Change in Financial Capability | study entry (pre-intervention), immediate post-intervention, 3 months post-intervention]
  The Financial Capability Scale measures one's knowledge, skills, and ability to manage financial resources effectively. It consists of 6 questions for which summed responses range between 0-8 points, with higher scores indicating greater feelings of financial capability.
Change in Financial Self-Sufficiency | study entry (pre-intervention), immediate post-intervention, 3 months post-intervention]
  The Financial Self-Sufficiency Scale assesses whether someone engages in sound money management activities such as comparison shopping, resisting impulse spending, living within their means, and balancing their bank account. This scale includes 6 items rated on a 4-point Likert scale ranging from "never true" to "always true" and summed for a total score potentially ranging from 6-24 points. Higher scores indicate greater financial self-sufficiency.
Change in Financial Literacy | study entry (pre-intervention), immediate post-intervention, 3 months post-intervention]
  The Financial Literacy Assessment tested knowledge of class content and included17 multiple-choice items with a 70% correct score considered passing in accordance with National Financial Educators Council guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Cook, Ph.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Department of Psychiatry, Chicago, Illinois, United States